CLINICAL TRIAL: NCT03199534
Title: A Prospective Cohort Trial of Pelvic Floor Chemodenervation in Patients Undergoing Physical Therapy for High Tone Pelvic Floor Dysfunction
Brief Title: A Trial of Pelvic Floor Chemodenervation in Patients Undergoing Physical Therapy for High Tone Pelvic Floor Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EvergreenHealth (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTPFD
Record Dates: First submitted 2017-06-13; First posted 2017-06-27 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Pelvic Pain; Dyspareunia; Pelvic Floor Dysfunction
Keywords: Pelvic Pain; Dyspareunia; Pelvic Floor Dysfunction; Pelvic Floor Physical Therapy; Chemodenervation; Botulinum Toxin A; Vaginismus
MeSH Terms: conditions — Pelvic Pain; Dyspareunia; Vaginismus | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Botulinum toxin A 50u (Experimental): Botulinum toxin A 50 unit injection
  Interventions: Drug: Botulinum toxin A 50u
- Botulinum toxin A 100u (Experimental): Botulinum toxin A 100 unit injection
  Interventions: Drug: Botulinum toxin A 100u
- Botulinum toxin A 150u (Experimental): Botulinum toxin A 150 unit injection
  Interventions: Drug: Botulinum toxin A 150u

INTERVENTIONS:
Drug: Botulinum toxin A 50u — Subject will receive injection of 50u Botulinum toxin A with local sedation as an office procedure.
  Other Names: BOTOX®; OnabotulinumtoxinA
  Arms: Botulinum toxin A 50u
Drug: Botulinum toxin A 100u — Subject will receive injection of 100u Botulinum toxin A in either the office or while anesthetized.
  Other Names: BOTOX®; OnabotulinumtoxinA
  Arms: Botulinum toxin A 100u
Drug: Botulinum toxin A 150u — Subject will receive injection of 150u Botulinum toxin A while anesthetized.
  Other Names: BOTOX®; OnabotulinumtoxinA
  Arms: Botulinum toxin A 150u

SUMMARY:
This study assesses whether the addition of chemodenervation to an established regimen of pelvic floor physical therapy for painful high tone pelvic floor dysfunction improves patients' objective and subjective outcomes. Study subjects will select one of three treatment approaches: injection of 50 units Botulinum toxin A with local sedation as an office procedure, injection of 100u BoNTA-cosmetic in either the office or while anesthetized, or injection of 150 units Botulinum toxin A while anesthetized.

DETAILED DESCRIPTION:
High-tone pelvic floor dysfunction is often a painful condition that can be associated with a number of female pelvic syndromes including childhood elimination disorders, idiopathic urinary retention, vaginismus, dyspareunia, pelvic pain, constipation, sport injuries, postoperative and bladder pain syndrome/interstitial cystitis. Following appropriate patient education about pelvic floor function, mainstays of therapy for high-tone pelvic floor dysfunction pelvic pain include pharmacotherapeutic agents and pelvic floor physical therapy. The investigators hypothesize that chemodenervation with Botulinum toxin A will offer a safe, efficacious intervention for women with high tone pelvic floor dysfunction that cannot be adequately treated with pelvic floor physical therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* >6 month history of pelvic pain or dyspareunia with high tone pelvic floor dysfunction on exam (pain with palpation of superficial transverse perineii, bulbocavernosus insertion to perineal/central tendon and/or levator ani complex/iliococcygeus)
* Women with male sexual partners
* History of undergoing pelvic floor physical therapy with internal manipulation including trigger point release as directed, with inability to meet goals of therapy despite appropriate pelvic floor physical therapy approach
* Able to read, write, and comprehend English sufficiently to offer informed consent

Exclusion Criteria:

* Presence of intact hymen, preventing internal manipulation during pelvic floor physical therapy
* Pregnancy at the time of injection
* Breast feeding at the time of injection
* History of Myasthenia Gravis, Amyotrophic Lateral Sclerosis, Lambert-Eaton syndrome, allergy to Botulinum toxin A, or other contraindication to Botulinum toxin A injection
* History of documented skin disorder of the vulva other than vaginal atrophy or lichen planus
* Prior pelvic radiation
* Stage II-IV pelvic organ prolapse
* Has had a pelvic floor Botulinum toxin A injection within the last 12 weeks
* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Pain Scale (Non-Menstrual Pelvic Pain) score | Baseline, Week 2, Month 3, Month 6, Month 9, Month 12
  This is a single question, "How severe is your pelvic pain at this time?"

SECONDARY OUTCOMES:
Visual Analog Pain Scale (Dyspareunia) | Baseline, Week 2, Month 3, Month 6, Month 9, Month 12
  This is a single question, "How severe was your pelvic pain the last time you had sexual intercourse?"
Patient Global Impression of Severity | Baseline, Week 2, Month 3, Month 6, Month 9, Month 12
  This questionnaire asks subjects to rate the severity of their pelvic pain symptoms. There are 4 choices to answer: 1 - Normal, no pain, 2 - Slightly more pain than normal, 3 - Significantly worse pain than normal, 4 - Severe pain.
Pelvic Floor Distress Inventory Questionnaire | Baseline, Week 2, Month 3, Month 6, Month 9, Month 12
  Subjects' rating on this 20-item questionnaire will be based on their bowel, bladder, and pelvic symptoms.
Female Sexual Function Index | Baseline, Week 2, Month 3, Month 6, Month 9, Month 12
  Subjects' rating on this 19-item questionnaire will be based on their sexual feelings and responses.
Patient Global Impression of Improvement | Week 2, Month 3, Month 6, Month 9, Month 12
  This questionnaire asks subjects to rate their current pelvic pain symptoms compared to before treatment. There are 7 choices to answer: 1 - very much better compared to before treatment, 2 - somewhat better compared to before treatment, 3 - slightly better compared to before treatment, 4 - no change compared to before treatment, 5 - slightly worse compared to before treatment, 6 - somewhat worse compared to before treatment, 7 - very much worse compared to before treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mia A. Swartz, MD, Principal Investigator — EvergreenHealth Urology & Urogynecology Care
Locations (1):
- EvergreenHealth Urology and Urogynecology Care, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.